CLINICAL TRIAL: NCT02071303
Title: Tramadol Versus Celecoxib for Reducing Pain Associated With Outpatient Hysteroscopy: A Randomized Double Blind Placebo-Controlled Trial
Brief Title: Tramadol Versus Celecoxib for Reducing Pain in Outpatient Hysteroscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer of Gynecology and Obstetrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Gany-124
Record Dates: First submitted 2014-02-23; First posted 2014-02-25 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2014-12

CONDITIONS: Pain
Keywords: Pain; Hysteroscopy; Tramadol; Celecoxib
MeSH Terms: conditions — Pain | interventions — Tramadol; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tramadol (Active Comparator): Women will receive Tramadol 100mg 1 hour before the procedure.
  Interventions: Drug: Tramadol
- Celecoxib (Active Comparator): Women will receive Celecoxib 200mg 1 hour before the procedure.
  Interventions: Drug: Celecoxib
- Placebo (Placebo Comparator): Women will receive a placebo 1 hour before the procedure.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tramadol — Tramadol 100mg will be given to 70 women before the procedure.
  Arms: Tramadol
Drug: Celecoxib — Celecoxib 200mg will be given to 70 women before the procedure.
  Arms: Celecoxib
Drug: Placebo — A placebo will be given to 70 women before the procedure.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effectiveness of Tramadol and Celecoxib in reducing pain during outpatient hysteroscopy. Women undergoing outpatient hysteroscopy in Cairo university will be divided into 3 groups, the first group will receive Tramadol 100 1 hour before the procedure, the second group will receive Celecoxib 200mg 1 hour before the procedure and the third will receive a placebo. Pain will be assessed by a visual analogue scale.

DETAILED DESCRIPTION:
Hysteroscopic examination is currently the most informative investigation for patients with abnormal uterine bleeding and infertility. Outpatient hysteroscopy involves the use of miniaturized endoscopic equipment to directly visualise the endometrial cavity, without the need of formal theatre facilities, general or regional anaesthesia.

Outpatient hysteroscopy is increasingly being used as a cost-effective alternative to in-patient hysteroscopy under general anaesthesia. Like other outpatient gynaecological procedures, however, it has the potential to cause pain severe enough for the procedure to be abandoned.

Several drugs have been used to reduce pain during the procedure. Celecoxib is a highly selective Cyclooxygenase-2 inhibitor (COX-2 inhibitor) whereas other Non-steroidal anti-inflammatory drugs (NSAIDS) like Ibuprofen, Diclofenac, and Naproxen inhibit both COX-1 and COX-2. COX-1 is the only isoenzyme found in platelets, and plays a role in the protection of the gastrointestinal mucosa, renal hemodynamics, and platelet thrombogenesis. In theory, this selectivity allows celecoxib and other COX-2 inhibitors to reduce inflammation and pain while minimizing gastrointestinal adverse drug reactions. COX-1 is involved in synthesis of prostaglandins and thromboxane, but COX-2 is only involved in the synthesis of prostaglandin. Therefore, inhibition of COX-2 inhibits only prostaglandin synthesis without affecting thromboxane, so offers no cardioprotective effects of nonselective NSAIDs .

Opioid analgesics are widely used for the control of moderate to severe pain. Tramadol hydrochloride, a synthetic opioid is an orally active, clinically effective centrally acting analgesic having a lower incidence of respiratory depression, cardiac depression, side effects on smooth muscle and abuse potential as compared to typical opioid agents.

The study will be conducted in the outpatient hysteroscopy clinic in Cairo university hospitals. All patients attending the outpatient hysteroscopy clinic will be invited to participate in the study. The invitation will include a clear full explanation of the study and patients will provide oral consent. Written informed consent is not needed since the procedure and intervention carries almost no risk to the patient and the patient will not receive anesthesia and will be fully conscious. Only patients consenting verbally to participate will be included in the trial.

Tramadol, celecoxib and placebo will be enclosed in sealed envelopes which will be numbered using computer generated random table. Neither the patient nor the physician will be aware of the drug used. 210 women will be categorized into 3 groups: Group I who will receive Tramadol 100mg (Trama SR®, Global Napi) orally 1 hour before the procedure, group II who will receive Celecoxib 200mg (Celebrex® 200, Pfizer) 1 hour before the procedure, and group III who will receive placebo acting as the control group.

Full history will be taken followed by general and local examination. The procedure will be done in the lithotomy position. Hysteroscopy will be done using a 5mm outer diameter continuous flow hysteroscope with a French working channel and a 30 degrees direction of view provided by Techno GmbH and CO. The hysteroscope will be introduced using the vaginoscopy technique, in which no speculum will be used. The cervix will be detected and the external os will be identified using the hysteroscope. The hysteroscope will be introduced in the uterine cavity. Saline will be used as the distension medium and the pressure will be set at 100mm Hg. The anterior wall, posterior wall and tubal ostea will be visualized, any polyps, adhesions septa, congenital malformations or submucous fibroids will be noted.

Base line characteristics and perception of pain will be compared.

ELIGIBILITY:
Inclusion Criteria:

* women referred to the outpatient hysteroscopy in Cairo university hospitals
* Consent to the procedure

Exclusion Criteria:

* Premenstrual patients
* Patients with missed periods
* Known cardiac disease
* Known gastritis or peptic ulcer
* Known allergy to Tramadol or Celecoxib

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Pain perception during the procedure | 10 minutes after starting the procedure.
  Pain will be assessed using a visual analogue scale 10 minutes after inserting the hysteroscope.

SECONDARY OUTCOMES:
Pain perception after the procedure | 30 minutes after the procedure.
  Pain will be assessed using a visual analogue scale 30 minutes after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: AbdelGany MA Hassan, MRCOG, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

REFERENCES:
- [Background] Sharma JB, Aruna J, Kumar P, Roy KK, Malhotra N, Kumar S. Comparison of efficacy of oral drotaverine plus mefenamic acid with paracervical block and with intravenous sedation for pain relief during hysteroscopy and endometrial biopsy. Indian J Med Sci. 2009 Jun;63(6):244-52. PMID 19602758
- [Background] van Dongen H, de Kroon CD, Jacobi CE, Trimbos JB, Jansen FW. Diagnostic hysteroscopy in abnormal uterine bleeding: a systematic review and meta-analysis. BJOG. 2007 Jun;114(6):664-75. doi: 10.1111/j.1471-0528.2007.01326.x. PMID 17516956
- [Background] O'Flynn H, Murphy LL, Ahmad G, Watson AJ. Pain relief in outpatient hysteroscopy: a survey of current UK clinical practice. Eur J Obstet Gynecol Reprod Biol. 2011 Jan;154(1):9-15. doi: 10.1016/j.ejogrb.2010.08.015. PMID 20926175
- [Background] Mathew ST, Devi S G, Prasanth VV, Vinod B. Efficacy and Safety of COX-2 Inhibitors in the Clinical Management of Arthritis: Mini Review. ISRN Pharmacol. 2011;2011:480291. doi: 10.5402/2011/480291. Epub 2011 May 17. PMID 22084715
- [Derived] Hassan A, Wahba A, Haggag H. Tramadol versus Celecoxib for reducing pain associated with outpatient hysteroscopy: a randomized double-blind placebo-controlled trial. Hum Reprod. 2016 Jan;31(1):60-6. doi: 10.1093/humrep/dev291. Epub 2015 Nov 29. PMID 26621854